CLINICAL TRIAL: NCT00439842
Title: HF Group Clinic Appointments: Rehospitalization Prevention
Brief Title: Self-Management and Care of Heart Failure With Group Clinics (SMAC-HF)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Carol Smith, RN, PhD, FAAN (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor-Investigator, Carol Smith, RN, PhD, FAAN, Professor, School of Nursing, University of Kansas Medical Center
Organization: University of Kansas Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1R01HL085397-05 (NIH); R01HL085397 (NIH)
Record Dates: First submitted 2007-02-22; First posted 2007-02-26 (Estimated); Last update posted 2015-04-17 (Estimated); Status verified 2015-04

CONDITIONS: Heart Failure, Congestive
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- HF group clinic appointments (Experimental): HF group clinic appointments Heart failure multidisciplinary group clinic appointments (Arm 1 - HFcareGroup) includes 6 teaching sessions with patients led by nurse practitioner.
  Interventions: Behavioral: Heart Failure Group Clinic Appointments
- Standard HF care (No Intervention): Standard HF care Standard heart failure education includes cardiologists instructions and hospital discharge information.

INTERVENTIONS:
Behavioral: Heart Failure Group Clinic Appointments — Self Management and Care of Heart Failure with Group Clinics (SMAC-HF)
  Other Names: HFcareGroup
  Arms: HF group clinic appointments

SUMMARY:
The purpose of this study is to help people with heart failure (HF) to manage their HF and to prevent rehospitalizations. Another purpose is to test the usefulness of clinical appointments and educational videotapes in teaching patients how to manage their HF.

It is proposed that the group clinic intervention (HFcareGroup)will reduce rehospitalization, depression, and improve problem solving related to heart failure symptoms.

DETAILED DESCRIPTION:
Aim 1 Hypothesis:

1. The time to the 1st composite endpoint (HF Rehospitalization/death) will be longer for HFcareGroup than standard care group at 12 months.
2. The HFcareGroup will have higher score than standard care on patient outcomes i.e. functional health status, quality of life, satisfaction with health care at 12 months.
3. Health Services Use will be lower in HFcareGroup than standard care group at 12 months.

Aim 2 Hypothesis:

1. The HFcareGroup will have higher score than standard care on patients' HF self-management i.e., self-care behaviors, participation with health care professionals in HF management and problem-solving, HF knowledge and preparedness for home care at 6 and 12 months.
2. A greater proportion of HFcareGroup vs standard care subjects will report clinical or symptoms of HF decompensation (e.g. specific weight gain, shortness of breath, edema, fatigue, tachycardia, and medication side effects) to their health care provider.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* speak English/Spanish
* receiving treatment for congestive heart failure
* receiving IV diuretics
* 2 or more HF symptoms
* be able to participate in follow up visits

Exclusion Criteria:

* primary right-sided heart failure
* HF transient & related to acute MI
* HF due to correctable cause
* being scheduled for coronary revascularization or any readmission
* receiving infusion for HF therapy within 2 weeks
* having co-morbidities, life expectancy < 12 months
* severe cognitive impairment
* D/C to nursing facilities or rehab unit
* Currently enrolled in an intervention study or HF management program
* being or planning to become pregnant within 12 months
* severe cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 2007-03; Primary Completion 2013-05 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
rehospitalization or death | 12 months

SECONDARY OUTCOMES:
HF self-management:problem-solving, self-care behaviors | 6 and 12 months
heart failure knowledge and preparedness for home care | 6 and 12 months
functional health status, quality of life, satisfaction with health care, health services use | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Carol Smith, PhD, RN, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

REFERENCES:
- [Derived] Piamjariyakul U, Shapiro AL, Wang K, Zulfikar R, Petitte T, Shafique S, Smith CE. Impact of Sleep Apnea, Daytime Sleepiness, Comorbidities, and Depression on Patients' Heart Failure Health Status. Clin Nurs Res. 2021 Nov;30(8):1222-1230. doi: 10.1177/10547738211015545. Epub 2021 May 12. PMID 33978519
- [Derived] Smith CE, Piamjariyakul U, Wick JA, Spertus JA, Russell C, Dalton KM, Elyachar A, Vacek JL, Reeder KM, Nazir N, Ellerbeck EF. Multidisciplinary group clinic appointments: the Self-Management and Care of Heart Failure (SMAC-HF) trial. Circ Heart Fail. 2014 Nov;7(6):888-94. doi: 10.1161/CIRCHEARTFAILURE.113.001246. Epub 2014 Sep 18. PMID 25236883